CLINICAL TRIAL: NCT03131934
Title: Immunotherapy With Tacrolimus Resistant EBV CTL for Lymphoproliferative Disease After Solid Organ Transplant
Acronym: ITREC
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Genetix Biotherapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL/16/0529
Record Dates: First submitted 2017-04-24; First posted 2017-04-27 (Actual); Last update posted 2024-05-17 (Actual); Status verified 2024-05

CONDITIONS: Post-transplant Lymphoproliferative Disease; Transplant-Related Hematologic Malignancy
MeSH Terms: interventions — Leukapheresis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Autologous EBV-CTL transduced with SFG-CNA12/SFG-CNA8 (Experimental): All patients will receive the autologous EBV CTL retrovirally transduced with with (a) a calcineurin mutant (CNA12) that confers resistance to tacrolimus and (b) a control calcineurin mutant (CNA8). For each patient two ATIMPs will be generated:
  * Autologous EBV-specific cytotoxic T-cells (CTL) transduced with the retroviral vector SFG-CNA12
  * Autologous EBV-specific cytotoxic T-cells (CTL) transduced with the control retroviral vector SFG-CNA8
  An equal dose (10x7/m2) of CNA12+ EBV CTL and CNA8+ EBV CTL will be administered intravenously on day 0.
  While awaiting ATIMP generation, patients may receive a single dose of Rituximab and other immunosuppressants (e.g. MMF) will be reduced, but tacrolimus will be maintained at therapeutic levels.
  Interventions: Biological: Autologous EBV-CTL transduced with vector SFG-CNA12; Biological: Autologous EBV-CTL transduced with control vector SFG-CNA8; Procedure: Leucapheresis

INTERVENTIONS:
Biological: Autologous EBV-CTL transduced with vector SFG-CNA12 — Autologous EBV-specific cytotoxic T-cells (CTL) transduced with the retroviral vector SFG-CNA12 conferring resistance to tacrolimus
Biological: Autologous EBV-CTL transduced with control vector SFG-CNA8 — Autologous EBV-specific cytotoxic T-cells (CTL) transduced with the control retroviral vector SFG-CNA8
Procedure: Leucapheresis — Patients will undergo an unstimulated leucapheresis to isolate the required immune cells to produce the EBV-CTLs

SUMMARY:
This is an open label, non-randomised, multicentre Phase I to determine the safety of tacrolimus-resistant autologous EBV-specific cytotoxic T-cells (EBV CTL) and compare their expansion/persistence with control EBV CTL in solid organ transplant patients with post-transplant lymphoproliferative disease (PTLD). Each patient will receive an infusion of two ATIMPs - autologous EBV CTL retrovirally transduced with (a) a calcineurin mutant (CNA12) that confers resistance to tacrolimus and (b) a control calcineurin mutant (CNA8).

DETAILED DESCRIPTION:
This is a multi-centre, non-randomised, open label Phase 1 clinical trial of Advanced Therapy Investigational Medicinal Products (ATIMPs) in adult and paediatric (age 1-70 years) solid organ transplant recipients with histologically proven B-lineage EBV+ post-transplant lymphoproliferative disease (PTLD).

The ATIMPs for this study are autologous EBV CTL transduced with the (a) the retroviral vector SFG-CNA12 encoding a calcineurin A mutant (CNA12) that confers resistance to tacrolimus and (b) the retroviral vector SFG-CNA8 encoding a control calcineurin A mutant (CNA8).

Following informed consent and registration to the trial, patients will undergo an unstimulated leucapheresis for generation of both ATIMPs. Patients will receive an equal dose of each ATIMP (10x7 CNA8+ or CNA12+ CTL/m2) which will be administered intravenously.

Other immunosuppressants (e.g. MMF) will be reduced, but tacrolimus will be maintained at therapeutic levels.The trial will evaluate the safety of the ATIMPs in organ transplant recipients developing EBV+ PTLD and compare the persistence and frequency of circulating CNA12 and CNA8 CTL in the peripheral blood.

Our hypothesis is that in the presence of ongoing immunosuppression with tacrolimus, CNA12 CTL will show preferential expansion and prolonged persistence compared with CNA8 CTL. If successful this will result in durable clearance of PTLD without the need to reduce tacrolimus, thus reducing the risk of graft rejection.

Patients will be followed up regularly during the interventional phase of the study until 1 year post EBV CTL infusion. During the long-term follow-up phase of the study (from 1-5 years post EBV CTL infusion) patients will be followed up annually.

ELIGIBILITY:
Inclusion Criteria:

1. Adult and paediatric (age 1-70 years) solid organ transplant recipients with histologically proven B-lineage EBV+ post-transplant lymphoproliferative disease (PTLD) either de novo or resistant to Rituximab
2. EBV viraemia at enrolment
3. On immunosuppression with tacrolimus
4. Agreement to have a pregnancy test and use of contraception for duration of trial (if applicable)
5. Written informed consent

Exclusion Criteria:

1. Fulminant disease
2. Requirement for supplemental oxygen
3. Burkitt's lymphoma/Mature B-acute lymphoblastic leukaemia with IgH-Myc rearrangement
4. T-lineage PTLD
5. Bilirubin > 3 x upper limit of normal
6. Creatinine > 3 x upper limit of normal
7. Active hepatitis B, C or HIV infection
8. Women who are pregnant or breast-feeding
9. ECOG performance score ≥ 4
10. Inability to tolerate leucapheresis

Ages: 1 Year to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2019-05-31 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2025-05-15 (Estimated)

PRIMARY OUTCOMES:
Toxicity at 6 weeks post infusion | 6 weeks
  Toxicity as assessed by NCI Common toxicity criteria within 6 weeks of infusion
Persistence and frequency of circulating EBV CTL | 12 months
  Persistence and frequency of circulating EBV CTL transduced with CNA12 compared with control vector CNA8 in the peripheral blood

SECONDARY OUTCOMES:
Disease response | 6 weeks
  Disease response at 6 weeks
Relapse rate | 2 years
  Relapse rate at 1 and 2 years
Disease free survival | 2 years
  Disease free survival at 1 and 2 yrs
Organ graft Rejection | 2 years
  Organ graft Rejection at 1 and 2 yrs

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Persis Amrolia, Principal Investigator — Great Ormond Street Hospital
Locations (2):
- United Kingdom (2):
  - Great Ormond Street Hospital, London
  - King's College Hospital, London

IPD SHARING:
Plan to Share IPD: Undecided